CLINICAL TRIAL: NCT03844477
Title: Quadratus Lumborum Block : Effect on Acute Pain and Quality of Recovery After Laparoscopic Adrenalectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We change the study protocal
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cui Xulei, Attending physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: cuixulei6
Record Dates: First submitted 2019-02-15; First posted 2019-02-18 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Pain Management; Nerve Block; Laparoscopic Adrenalectomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-injection QLB(quadratus lumborum block) (Experimental): Single-injection of QLB with local anesthetic is given preoperatively
  Interventions: Procedure: single-injection QLB(quadratus lumborum block)
- Placebo control (Placebo Comparator): Single-injection of QLB with NS is given preoperatively
  Interventions: Procedure: Placebo control

INTERVENTIONS:
Procedure: single-injection QLB(quadratus lumborum block) — Inject 0.4ml/kg 0.5% ropivacaine between quadratus lumborum and psoas major without continuous local infusion
  Device: Ultrasound Scanner The curved (C1-5) probe of Ultrasound Scanner is used for scan
  Device: PAJUNK StimuLong Drug: single dose ropivacaine 0.4ml/kg 0.5% ropivacaine given immediately after the correct position of the tip of the needle has been verified.
  Arms: single-injection QLB(quadratus lumborum block)
Procedure: Placebo control — Inject 0.4ml/kg saline between quadratus lumborum and psoas major without continuous local infusion
  Device: Ultrasound Scanner The curved (C1-5) probe of Ultrasound Scanner is used for scan
  Device: PAJUNK StimuLong Drug: single dose 0.4ml/kg 0.9% NS. given immediately after the correct position of the tip of the needle has been verified.
  Arms: Placebo control

SUMMARY:
This prospective, randomized ,control study aims to compare the analgesic effect,quality of recovery, length of hospital stay ,et al. between single-injection QLB(quadratus lumborum block)+general anesthesia (GA) and general anesthesia (GA) alone in patients undergoing laparoscopic adrenalectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 yrs
* American Society of Anesthesiologists physical statusⅠ-Ⅲ
* Undergo laparoscopic adrenalectomy
* Informed consent

Exclusion Criteria:

* A known allergy to the drugs being used
* Coagulopathy, on anticoagulants
* Analgesics intake, history of substance abuse
* Participating in the investigation of another experimental agent
* Inability to properly describe postoperative pain to investigators (eg, language barrier, neuropsychiatric disorder)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-16 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
pain numeric rating scale (NRS, 0-10)pain score at activity at 12 hours after surgery | At 12hours after the surgery

SECONDARY OUTCOMES:
The pain scores at rest determined by the numeric rating scale (NRS, 0-10) | At 2,4, 8, 12,24 ,48,72hours after the surgery
incidence of postoperative nausea and vomiting (PONV) | within 24 postoperative hours
ambulation time | within5 days after surgery
time of restart anal exhaust | within 5 days after surgery
Postoperative length of hospital stay | up to2 weeks after surgery
patient's satisfaction with anesthesia and analgesia | 48 hours after surgery
  use the Chinese version Bauer questionnaire to assess the patient satisfaction with anesthesia and analgesia
The pain scores at activity determined by the numeric rating scale (NRS, 0-10) | At 2,4, 8, 24 ,48,72hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xulei CUI, md, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No